CLINICAL TRIAL: NCT00026052
Title: An Investigation of the Antidepressant Efficacy of an Antiglutamatergic Agent With Neurotrophic Properties in Major Depression
Brief Title: Riluzole to Treat Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020034; 02-M-0034
Record Dates: First submitted 2001-11-08; First posted 2001-11-09 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Depression
Keywords: Riluzole; Neuroprotective; Open-Label Study; Glutamate Dysfunction; Unipolar Depression; Antidepressant; Depression; Major Depression
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major | interventions — Riluzole

INTERVENTIONS:
Drug: riluzole

SUMMARY:
This study will examine the safety and effectiveness of the drug riluzole (Rilutek® (Registered Trademark)) for short-term treatment of depression symptoms, such as depressed mood, psychomotor retardation, and excessive sleeping. Despite the availability of a wide range of antidepressant drugs, studies indicate that 30 to 40 percent of patients with major depression do not respond to first-line antidepressant treatment with drugs such as fluoxetine, upropion, venlafaxine and others. Riluzole, which is approved by the Food and Drug Administration (FDA) for amyotrophic lateral sclerosis (ALS), causes chemical changes in the brain that may also have antidepressant properties.

Patients between 18 and 70 years of age with major depressive disorder without psychotic features may be eligible for this 2-stage 7-week study. Candidates will be screened with a medical history and physical examination, including an electrocardiogram (EKG), blood and urine tests, and a psychiatric evaluation. A

blood or urine sample will be tested for illegal drugs.Women of childbearing potential will have a pregnancy test.

Participants will complete stage 1 of the study, which lasts 1 week, and may then continue with stage 2 for an additional 6 weeks. At the start of the study, patients will be tapered off all psychiatric medicines and will begin treatment with a placebo (a sugar pill formulated to look like the active drug). At some point, they will be switched from placebo to riluzole. In addition, participants will undergo the following procedures:

* Physical examination and electrocardiograms (EKG) at the beginning and end of the study, with vital signs (temperature, blood pressure and heart rate) checked daily
* Weekly 1-hour interviews consisting of psychiatric and psychomotor rating scales to assess treatment response
* Weekly blood tests to measure blood levels of riluzole and evaluate drug side effects

At the end of the study, participants' psychiatric status will be reassessed and appropriate long-term psychiatric treatment arranged.

Patients, ages 18 to 70 with a diagnosis of major depression without psychotic features, will in this pilot study (single arm, single blind) receive riluzole (50-200 mg/day) for a period of 6 weeks. Acute efficacy will be determined by demonstrating a greater response rate using specified criteria.

Approximately 25 patients will enter the study to obtain 22 subjects who complete the 6 weeks of acute riluzole treatment. Therefore, if 7/22 patients or greater have greater than 50% improvement on the primary efficacy measure, then based on statistically guidelines from the Optimal Two Stage Design for Clinical Trials, a controlled trial would be indicated to scientifically confirm the signal observed in the single arm trial.

DETAILED DESCRIPTION:
Major affective disorders are common, severe, chronic and often life-threatening illnesses. Major depression contributes to significant morbidity and mortality. Impairment in physical and social functioning resulting from depression can be just as severe as other chronic medical illnesses. Suicide is the cause of death in 10-20% of individuals with either bipolar or recurrent depressive disorders.

Despite the availability of a wide range of antidepressant drugs, clinical trials indicate that 30% to 40% of patients with major depression fail to respond to first-line antidepressant treatment, despite adequate dosage, duration, and compliance. Thus, there is a clear need to develop novel and improved therapeutics for unipolar and bipolar depression. Recent preclinical studies suggest that antidepressants may exert delayed indirect effects on the glutamatergic system. Furthermore, a growing body of data suggests that mood disorders are associated with regional volumetric reductions, and cell loss and atrophy. It is thus noteworthy that lamotrigine, which, among other effects reduces glutamate release, has antidepressant effects, and a pilot study has suggested that NMDA antagonists may have antidepressant effects. Together, this data suggests that the glutamatergic system may play a role in the pathophysiology and treatment of depression, and that agents, which more directly reduce glutamatergic neurotransmission, may represent a novel class of antidepressants.

Riluzole, an agent that is Food and Drug Administration-approved for Amyotrophic Lateral Sclerosis has significant antiglutamatergic and neuroprotective properties, may prove to have antidepressant properties in depressed patients. In this study, we propose to investigate the potential antidepressant efficacy of riluzole, an agent which reduces glutamatergic throughput via inhibition of its release, which also exerts robus neurotrophic effects.

This is a 6-week single-arm, single-blind study that will examine the efficacy and safety of riluzole in patients with major depression without psychotic features.

The study has two Study Periods. Study Period I is the washout phase that will last 7 days. Study Period II is a monotherapy 6-week acute treatment phase in which the efficacy and tolerability of riluzole is compared to baseline.

Patients, ages 18 to 60 with a diagnosis of major depression without psychotic features, will in this pilot study (single arm, single-blind) receive riluzole (50-200 mg/day) for a period of 6 weeks. Acute efficacy will be determined by demonstrating a greater response rate using specified criteria.

Approximately 25 patients will enter the study to obtain 22 subjects who complete the 6 weeks of acute riluzole treatment. Therefore if 7/22 patients or greater have greater than 50% improvement on the primary efficacy measure, then based on statistically guidelines from the Optimal Two Stage Design for Clinical Trials, a controlled trial would be indicated to scientifically confirm the signal observed in the single arm trial.

ELIGIBILITY:
INCLUSION CRITERIA

Male or female subjects, 18 to 70 years of age will be eligible.

Female subjects of childbearing potential must be using a medically accepted means of contraception.

Each subject must have a level of understanding sufficient to agree to all required tests and examinations.

Each subject must understand the nature of the study and must sign an informed consent document.

Subjects must fulfill the criteria for major depression, recurrent without psychotic features as defined in DSM-IV (296.32, 296.33) based on clinical assessment and confirmed by structured diagnostic interview SCID-P.

Subjects must have an initial score at Visit 1 and Visit 2 of at least 20 on the MADRS.

Subjects must not have a decrease in the total score of MADRS of greater than or equal 20% during washout (between Visits 1 and 2).

Subjects must have experienced, in the opinion of the investigator, at least one prior major depressive episode as defined in DSM-IV (not including the current major depressive episode).

Subjects must have had at least one adequate antidepressant trial (SSRI, bupropion, or venlafaxine) during an episode of major depression (Thase and Rush, 1995; Thase et al., 2000).

Subjects with current major depressive episode of no more than 24 months will be eligible.

EXCLUSION CRITERIA

Presence of psychotic features.

Participate in a clinical trial of another investigational drug within 1 month (30 days) prior to study entry (Visit 1).

Female subjects who are either pregnant or nursing.

Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.

Subjects with uncorrected hypothyroidism or hyperthyroidism.

Abnormal levels of serum transaminases (ALT/SGPT; AST/SGOT), current or past blood dyscrasia.

Documented history of hypersensitivity or intolerance to riluzole.

DSM-IV substance abuse or dependence within the past 90 days.

Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections prior to Visit 2.

Treatment with a reversible MAOI, guanethidine, or guanadrel within 1 week or with fluoxetine within 3 weeks prior to Visit 2.

Treatment with any other concomitant medication with primarily CNS activity, other than specified in Appendix A.

Treatment with clozapine or ECT within 12 weeks prior to Visit 2.

Current diagnosis of schizophrenia or other psychotic disorder as defined in the DSM-IV will be excluded.

Judged clinically to be at serious suicidal risk, with a score of 3 or more on item 3 of the HAMD will be excluded.

Patients will not be allowed to receive structured psychotherapy during the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31
Dates: Start 2001-11; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Aronowski J, Strong R, Grotta JC. Combined neuroprotection and reperfusion therapy for stroke. Effect of lubeluzole and diaspirin cross-linked hemoglobin in experimental focal ischemia. Stroke. 1996 Sep;27(9):1571-6; discussion 1576-7. doi: 10.1161/01.str.27.9.1571. PMID 8784132
- [Background] Altamura CA, Mauri MC, Ferrara A, Moro AR, D'Andrea G, Zamberlan F. Plasma and platelet excitatory amino acids in psychiatric disorders. Am J Psychiatry. 1993 Nov;150(11):1731-3. doi: 10.1176/ajp.150.11.1731. PMID 8214185
- [Background] Abe K, Aoki M, Kawagoe J, Yoshida T, Hattori A, Kogure K, Itoyama Y. Ischemic delayed neuronal death. A mitochondrial hypothesis. Stroke. 1995 Aug;26(8):1478-89. doi: 10.1161/01.str.26.8.1478. PMID 7631357